CLINICAL TRIAL: NCT05737914
Title: Bilateral Endoscopic Thoracic T3 Sympathectomy Versus T3 Radiofrequency Ablation for Treatment of Primary Palmar Hyperhidrosis
Brief Title: Bilateral Endoscopic Thoracic T3 Sympathectomy Versus T3 Radiofrequency Ablation for Primary Palmar Hyperhidrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R 36 /2018
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Primary Palmar Hyperhydrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic thoracic T3 sympathectomy (Active Comparator)
  Interventions: Procedure: Endoscopic thoracic T3 sympathectomy
- ThoracicT3 radiofrequency ablation (Active Comparator)
  Interventions: Procedure: ThoracicT3 radiofrequency ablation

INTERVENTIONS:
Procedure: Endoscopic thoracic T3 sympathectomy — Interruption of intrathoracic sympathetic neural pathway surgically to treat hyperhidrosis by using video - thoracoscopy
  Arms: Endoscopic thoracic T3 sympathectomy
Procedure: ThoracicT3 radiofrequency ablation — radiofrequency ablation at third thoracic spine it may be a good option for treatment of primary hyperhidrosis.
  Arms: ThoracicT3 radiofrequency ablation

SUMMARY:
Primary hyperhidrosis disease is characterized by much more sweating above the needs for thermoregulation, which is worsen by increased temperature and emotional factors it can be seen in the palms of the hands, soles of the feet/ face and so on.

Hyperhidrosis usually starts since childhood and continuous throughout life aggravated by emotional stress or by high environmental temperature.

Many lines of treatment were tried such as anticholinergic drug, physiotherapy. Endoscope thoracic sympathectomy and radio frequency with phenol injection.

DETAILED DESCRIPTION:
Interruption of intrathoracic sympathetic neural pathway surgically to treat hyperhidrosis by using video - thoracoscopy which has lead to explosion of minimally invasive technique for this issue. It's safe procedure and success rate in about 95% so it's result in this disease are rewarding.

Other technique will be studied in this current study is radiofrequency ablation it may be a good option for treatment of primary hyperhidrosis. When endoscope is not allowed.

An early outcome is our primary target for comparing the two different techniques.

Treatment with radiofrequency can benefit patients specially young one because a lot of them refuse endoscopic sympathectomy with its special anesthetic consideration as one lung ventilation and sometimes patient left with intercostal tube for some days so it's considered difficult procedure and much more easy is radiofrequency but alone the results is not satisfactory so in this clinical trial endoscopic sympathectomy will be compared with radiofrequency ablation regarding to the early outcome for the two procedure in this clinical trial interruption of sympathetic chain was chosen at the level of T3 because at this level interruption involve only the sympathetic chain without any ganglion damage or compensatory sweating which was seen when the interruption of the level of T4.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary palmar hyperhydrosis.
* Patients with American society classification 1 and 2.

Exclusion Criteria:

* Patient refusal.
* Previous sympathectomy either endoscopic or by radiofrequency.
* Previous sternotomy operation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
success rate | one week after surgery
  measured by the hyperhidrosis disease severity score. A score of 1 or 2 was classified as mild or moderate hyperhidrosis and a score of 3 or 4 was classified as severe hyperhidrosis.
success rate | one month after surgery
  measured by the hyperhidrosis disease severity score. A score of 1 or 2 was classified as mild or moderate hyperhidrosis and a score of 3 or 4 was classified as severe hyperhidrosis.

SECONDARY OUTCOMES:
compensatory sweating | one week after surgery
  detected by sweating of chest, abdomen, back, head and neck
compensatory sweating | one month after surgery
  detected by sweating of chest, abdomen, back, head and neck
number of patients develope pneumothorax | immediately after surgery
  detected by chest x ray
recurrence of sweating | one week after surgery
  measured by the hyperhidrosis disease severity score. A score of 1 or 2 was classified as mild or moderate hyperhidrosis and a score of 3 or 4 was classified as severe hyperhidrosis.
recurrence of sweating | one month after surgery
  measured by the hyperhidrosis disease severity score. A score of 1 or 2 was classified as mild or moderate hyperhidrosis and a score of 3 or 4 was classified as severe hyperhidrosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No